CLINICAL TRIAL: NCT01953341
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 333 in Healthy Subjects and Subjects With Migraines.
Brief Title: Single-Ascending Dose Study of AMG 333 in Healthy Subjects and Subjects With Migraines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20130102
Record Dates: First submitted 2013-09-26; First posted 2013-09-30 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — AMG 333

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 333 (Experimental): Subjects will receive a single oral dose of AMG 333 .
  Interventions: Drug: AMG 333
- Placebo (Placebo Comparator): Subjects will receive a single oral dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 333 — Oral administration available in varying dose strength.
  Arms: AMG 333
Drug: Placebo — Placebo containing no active drug
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine whether AMG 333 is safe and well tolerated in healthy subjects and subjects with migraines. As part of the secondary objectives, this study will characterize the pharmacokinetic (PK) profile of AMG 333, as well as characterize the effect of AMG 333 on the cold pressor test (CPT)-induced increase in blood pressure after single oral doses in healthy subjects and subjects with migraines

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, ascending single-dose study evaluating AMG 333 in healthy subjects and subjects with migraines. The study will consist of 8 cohorts: 7 cohorts of healthy subjects and 1 cohort of subjects with migraines. For cohorts 1 to 7, 8 subjects each will be enrolled, and subjects will be randomized such that 6 subjects will receive AMG 333 and 2 subjects will receive placebo (3:1 ratio). In cohort 8, up to 24 subjects with migraines will be enrolled, depending on enrollment rate and emerging safety and tolerability data. These migraine subjects will be randomized to receive AMG 333 or placebo in a crossover fashion. Both healthy and migraine subjects will be monitored in house for 4 days then allowed to return home for the remainder of the 14 day observation period. Both healthy and migraine subjects will keep headache diaries.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects with or without migraines ≥18 and ≤55 years of age at the time of screening, with no history or evidence of clinically relevant medical disorders as determined by the investigator in consultation with the Amgen physician.

Exclusion Criteria:

* History or evidence of a clinically significant disorder, condition, or disease that, in the opinion of the investigator and Amgen physician, would significantly impair pain perception (eg, history of stroke, history of neuropathy) or interfere with evaluation, procedures, or study completion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Primary | Up to 29 days
  Treatment-emergent adverse events, including changes in vital signs, 12-lead ECGs, clinical laboratory safety tests, and physical and neurological assessments
Primary | Up to 29 days
  Headache assessment as measured by the occurrence of moderate-to-severe headache within 36 hours of treatment, as well as number of moderate-to-severe headaches within 4 days of dosing

SECONDARY OUTCOMES:
Secondary Outcome Measures | Up to 29 Days
  Time to maximum concentration [Tmax])
Secondary | Up to 29 days
  Change in systolic and diastolic blood pressure in response to Cold Pressor Test (CPT)
Secondary Outcome Measures | Up to 29 Days
  Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration [AUClast]
Secondary Outcome Measures | Up to 29 Days
  Area under the concentration-time curve from time 0 extrapolated to infinity [AUCinf], maximum observed concentration [Cmax], and T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Salt Lake City, Utah, United States

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com